CLINICAL TRIAL: NCT01747239
Title: Cabazitaxel in Platinum Refractory Ovarian Cancer. A Phase II Trial
Brief Title: Cabazitaxel in Platinum Refractory Ovarian Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Too low inclusion rate. Only 4 patients included over 16 months
Sponsor: Vejle Hospital (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TaxOvar
Record Dates: First submitted 2012-12-06; First posted 2012-12-11 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Ovarian Cancer
Keywords: Ovarian cancer; Platinum refractory
MeSH Terms: conditions — Ovarian Neoplasms | interventions — cabazitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cabazitaxel (Experimental): 25 mg/m2 IV every three weeks
  Interventions: Drug: Cabazitaxel

INTERVENTIONS:
Drug: Cabazitaxel — 25 mg/m2 IV every three weeks

SUMMARY:
Ovarian cancer patients are considered platinum refractory if their disease worsens during primary platinum treatment or if they have no effect of the treatment. This constitutes a major therapeutic problem and new treatment approaches are highly needed.

Cabazitaxel (Jevtana®) is a new taxane with effect in breast and prostatic cancer. In both tumors it has effect in patients refractory to taxotere. Consequently, it could be anticipated that cabazitaxel may have an effect in platinum refractory ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed epithelial, primary fallopian or primary peritoneal cancer. Stages I-IV.
* Patients with refractory disease defined as progression or no change during primary treatment, as evaluated after 3 and/or 6 cycles of platinum/paclitaxel. Prior to inclusion, patients must have received platinum and paclitaxel as combination treatment.
* Measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 or evaluable by Gynecologic Cancer Interest Group (GCIG) cancer antigen 125 (CA-125) criteria.
* Age ≥ 18 years.
* Performance stage 0-2.
* Adequate bone marrow function, liver function, renal function, and coagulation parameters (within 7 days prior to inclusion):

  1. Neutrophils (ANC) ≥ 1.5 x 10^9/l
  2. Platelet count ≥ 100 x 10^9/l
  3. Serum bilirubin ≤ 1.0 x upper limit of normal (ULN)
  4. Serum transaminase ≤ 2.5 x ULN
  5. Serum creatinine ≤ 1.5 ULN. If creatinine 1.0 - 1.5 x ULN, creatinine clearance will be calculated according to the Chronic Kidney Disease Epidemiology Collaboration formula (CKD-EPI)and patients with creatinine clearance <60 mL/min should be excluded
* Written informed consent.

Exclusion Criteria:

* History of severe hypersensitivity reaction (≥grade 3) to taxol.
* History of severe hypersensitivity reaction (≥grade 3) to polysorbate 80 containing drugs.
* Concurrent or planned treatment with strong inhibitors or strong inducers of cytochrome P4503A4/5 (a one week wash-out period is necessary for patients who are already on these treatments).
* Neuropathy grade ≥ 2.
* Pregnant or breast-feeding patients. For fertile women a negative pregnancy test at screening is mandatory.
* Fertile patients not willing to use effective methods of contraception during treatment and for 6 months after the end of treatment.
* Other malignant diseases within 5 years prior to inclusion in the study, except basal cell or squamous cell carcinoma of the skin and cervical carcinoma-in-situ.
* Other experimental therapy or participation in another clinical trial within 28 days prior to treatment initiation.
* History of any chronic medical or psychiatric condition or laboratory abnormality that is not medically controlled or in the opinion of the investigator may increase the risks associated with study drug administration. (e.g. diabetes, cardiac diseases, hypertension, renal, thyroid or liver disease).
* Vaccination with yellow fever vaccine or any live attenuated vaccine during the treatment.
* Treatment with disulfiram (antabuse)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2013-01; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Rate of response to cabazitaxel | Every 9 weeks up to two years
  Response must be confirmed by a second CT scan 4-6 weeks after first response by CT scan

SECONDARY OUTCOMES:
Progression free survival | Every three months until progression or death, up to three years
Overall survival | Every 3 months up to three years

CONTACTS AND LOCATIONS:
Overall Officials: Anders Jakobsen, DMSc, Study Chair — Vejle Hospital; Christine V Madsen, MD, Principal Investigator — Vejle Hospital
Locations (4):
- Denmark (4):
  - Department of Oncology, Aalborg Hospital, Aalborg
  - Herlev Hospital, Herlev
  - Department of Oncology, Odense University Hospital, Odense
  - Department of Oncology, Vejle Hospital, Vejle